CLINICAL TRIAL: NCT06372509
Title: A Proteomic Analysis for Understanding the Link Between Migraine and Cardiovascular Disease
Acronym: PMCD
Status: Recruiting | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: IRCCS Policlinico S. Donato (Other)
Responsible Party: Sponsor
Other Study IDs: L2-070
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Migraine; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Migraine Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample will be used for a targeted proteomic assessment of proteins relevant in CVD, inflammation, immune response and neurological disorders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with migraine: Consecutive patients admitted for non coronary disease, will follow their clinical pathway. They will be classified into symptomatic for migraine with aura (group 1, N=45) and free from migraine (N=45) and will be enrolled in the study.
- Patients w/o migraine: Consecutive patients admitted for non coronary disease, will follow their clinical pathway. They will be classified into free from migraine (group 2, N=45) and will be enrolled in the study.

SUMMARY:
This is a multicenter, prospective observational study. Will be collecting data from 90 consecutive patients (aged 25- 60 years ) with and without migraine admitted at our Hospital. Primary aim of the study will be to assess the correlation between migraine and proteomic profiling of plasma and their possible correlation with known cardio and cerebrovascular disease and Cardiovascular (CV) risk factors.

DETAILED DESCRIPTION:
Ninety consecutive patients hospitalized for noncoronary artery disease will follow their clinical course. They will be classified into symptomatic for migraine with aura (N=45) and migraine free (N=45) and will be enrolled in the study. Patients will be screened for migraine characteristics and a comprehensive clinical analysis, including sex-related cardiovascular risk factors, will be collected. To achieve the study objective, blood will be drawn to do targeted proteomic evaluation of proteins relevant to Cardiovascular disease (CVD), inflammation, immune response, and neurological disorders, in order to compare the profile of migraine patients with that obtained in patients without migraine.

ELIGIBILITY:
Inclusion Criteria:

* Age >25 years and > 60 years
* Signed patient informed consent form (ICF)
* Non-coronary disease

Exclusion Criteria:

* Age < 25 years and > 60 years
* Acute myocardial infarction (MI)
* Chronic kidney disease: glomerular filtration rate (GFR) < 30 ml/min
* Severe mitral or aortic valvular disease
* Acute heart failure
* Reduced left ventricular (LV) function (Ejection Fraction < 35%)
* Atrial Fibrillation

Ages: 25 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Consecutive patients admitted for non coronary disease, will follow their clinical pathway. They will be classified into symptomatic for migraine with aura (N=45) and free from migraine (N=45) and will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between migraine and proteomic profiling of plasma | October 2025
  A blood sample will be obtained to perform a targeted proteomic assessment of proteins relevant in CVD, inflammation, immune response and neurological disorders in order to compare migraineurs patients profile with the one obtained in migraine-free patients

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Milan, Milan, Italy